CLINICAL TRIAL: NCT05160428
Title: New or Flare of Musculoskeletal Rheumatic Diseases After Different COVID-19 Vaccines: Multicentre Study
Brief Title: Post Covid-19 Vaccination Development or Flare of ARD
Acronym: PoCov-ARD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mervat Eissa, Associate Professor, Cairo University
Other Study IDs: Post Covid Vaccination ARD
Record Dates: First submitted 2021-12-14; First posted 2021-12-16 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; Vaccination; Infection; Rheumatic Diseases
MeSH Terms: conditions — COVID-19; Infections; Rheumatic Diseases | interventions — heterologous prime boost COVID-19 vaccination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: COVID-19 vaccination — different types of covid-19 vaccinations.

SUMMARY:
Many patients develop autoimmune diseases after covid-19 vaccination, whether related to the vaccination or not, is still under study. This study will describe potential flare of ARD after COVID-19 vaccination, whether it leads to activity or new MSK manifestations development.

DETAILED DESCRIPTION:
-In this study: patients with known diagnosed rheumatic diseases who are vaccinated (one or full doses) of any type of COVID-19 vaccines will be enrolled. new ARD and prevalence of different MSK manifestations after covid-19 vaccinations also will be reported. The prevalence of flare of ARD after covid-19 vaccinations will be dteremined. Also we will compare between different types and doses of covid-19 vaccinations in inducing ARD or flares.

Study Design: Cross sectional study Target population: any patient with pre-existing received any vaccination against covid-19 visiting rheumatology outpatient clinic.

-any patient develops MSK manifestations after covid-19 vaccination. The disease activity sataus will be measured according to the type of rheumatic disease. For RA , disease activity score28 will be used, in lupus: SLEDAI, in Behcet : BDCAF, in SpA: BASDAI.

ELIGIBILITY:
Inclusion Criteria:

Age above 18 years Vaccinated against covid-19 (one dose or fully vaccinated)

Exclusion Criteria:

Receiving other vaccine e.g influenza Less than 18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligibility Criteria:
  Patients above 18 years old having MRD manifestations vaccinated against covid-19.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
-Prevalence of new ARD after covid-19 vaccinations | 3 moths
  any ARD
prevalence of flare of ARD after covid-19 vaccinations | 3 months
  flare of any manifestations of the disease

SECONDARY OUTCOMES:
Prevalence of non-specific MSK symptoms after Covid-19 vaccine. | 3 months
  any MSK symptoms
Correlation of the MSK to the 1st and 2nd Covid vaccine dose | 3 months
  Correlation of the MSK to the 1st and 2nd Covid vaccine dose
comparison between different type of covid-19 vaccine in inducing ARD or flare up. | 3 months
  any type of flare
disease activity status in the patients who developed the ARD symptoms before and after the vaccine. | 3 months
  activity assessed by disease activity scores
Any correlation between the appearance of MSK symptoms and the patient's medications | 3 months
  current medications

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abuzaid, MD, Principal Investigator — Tanta University
Locations (1):
- Kasr Alainy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided